CLINICAL TRIAL: NCT01903902
Title: The Efficacy and Safety of Paclitaxel-eluting SeQuent Please Drug-Eluting Balloon for Treatment of lesiOns in Native smalL coronarY Arteries (DEB-ONLY)
Brief Title: Efficacy and Safety of Paclitaxel-eluting Balloon for Treatment of Lesions in Native Small Coronary Arteries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Inje University (Other); Chonnam National University Hospital (Other); Ulsan University Hospital (Other); Jeju National University Hospital (Other); Daegu Catholic University Medical Center (Other); Chungbuk National University (Other); Dankook University (Other); The Catholic University of Korea (Other); Kwandong University Myongji Hospital (Unknown); Kosin University Gospel Hospital (Other); Keimyung University Dongsan Medical Center (Other); Soonchunhyang University Hospital (Other); National Health Insurance Service Ilsan Hospital (Other); Saint Carollo General Hospital (Unknown); Chuncheon Sacred Heart Hospital (Other); Sejong General Hospital (Other); Cheju Halla General Hospital (Other); Wonkwang University (Other); Konyang University Hospital (Other); Gangnam Severance Hospital (Other); Hallym University Medical Center (Other); Chonbuk National University Hospital (Other); Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Woong Chol Kang, Associate Professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEB-ONLY
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Balloon angioplasty; Drug-eluting balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug-eluting balloon (Experimental): Balloon angioplasty using paclitaxel-eluting SeQuent Please drug-eluting balloon in native small coronary artery (vessel diameter > 2.25 mm and ≤ 2.75 mm)
  Interventions: Device: SeQuent® Please Drug-eluting balloon

INTERVENTIONS:
Device: SeQuent® Please Drug-eluting balloon — Balloon angioplasty using paclitaxel-eluting balloon (SeQuent® Please) will be done in native small coronary artery (vessel diameter ≥ 2.25 mm and ≤ 2.75 mm, and lesion length < 25 mm), if residual stenosis is ≤ 30% and there are no dissection of classification C and over which disturbed blood flow after plain balloon angioplasty.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of paclitaxel-eluting balloon (SeQuent® Please) for treatment of lesions in native small coronary arteries.

DETAILED DESCRIPTION:
Drug-eluting balloon (DEB) have emerged as a potential alternative to overcome the limitations of drug-eluting stents such as restenosis or stent thrombosis.

DEB angioplasty is proven to be effective clinically for the treatment of in-stent restenosis. However, DEB for de novo lesions, especially in small vessels is less studied.

The purpose of this study is to evaluate the efficacy and safety of paclitaxel-eluting balloon (SeQuent® Please) for treatment of lesions in native small coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Patients who are appropriate for percutaneous coronary intervention using drug-eluting balloon in native small coronary artery (vessel diameter ≥ 2.25 mm and ≤ 2.75 mm, lesion length < 25 mm)
* Informed consent

Exclusion Criteria:

* Chronic total obstruction lesion
* Severe calcified lesion
* Left main coronary lesion
* Lesion having intravascular thrombus
* Shock status from any cause including cardiogenic shock
* Left ventricular ejection fraction < 30%
* Need for coronary artery bypass surgery
* Allergic reaction for paclitaxel
* Severe allergic for contrast agent (Visipaque) or statin
* Pregnancy, breastfeeding or Expectation for pregnancy in women of childbearing age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Late loss | 9±1 months
  Late loss of the target lesion at the follow-up (9±1 months) quantitative coronary
Binary restenosis rate | 9±1 months
  Restenosis rate of the target lesion at the follow-up quantitative coronary angiography

SECONDARY OUTCOMES:
Neointimal hyperplasia | 9±1 months
  Neointimal hyperplasia of the target lesion at the follow-up intravascular ultrasound (IVUS) or optical coherence tomography (OCT) exam
Clinical outcomes | 9±1 months
  Clinical outcomes including death, myocardial infarct, target lesion revascularization, stent thrombosis within the target lesion

CONTACTS AND LOCATIONS:
Overall Officials: Woong Chul Kang, M.D., Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea